CLINICAL TRIAL: NCT03140865
Title: Wake Forest Alzheimer's Disease Clinical Core
Acronym: ADCC
Status: Recruiting | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB00025540; 40010560 (Other: National Institute on Aging)
Record Dates: First submitted 2014-12-19; First posted 2017-05-04 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-04

CONDITIONS: Alzheimer's Disease; Mild Cognitive Impairment; Prediabetic State
Keywords: Alzheimer's; observational; prediabetes; mild cognitive impairment
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction; Prediabetic State

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Blood collection for routine laboratory tests (hemoglobin A1c, CBC, BMP 8, lipid panel, TSH, Vitamin B12, insulin, and coagulation). Blood will also be drawn for genotyping and determining ApoE status as well as stored for future assays.
  CSF will be collected on a subset of participants and used to analyze amyloid beta, t-tau, p-tau, and stored for future assays.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cognitively Normal: This group will include 300 healthy volunteers with no apparent memory problems. Participants will complete an assessment at enrollment and once per year for the following 5 years. In addition to memory assessments at baseline and year 4, participants will have a brain MRI, OGTT A reliable study partner will need to attend the visits or be available via telephone to complete study interviews.
- Mild Cognitive Impairment: This group will include 400 volunteers who have mild memory problems that are observed during cognitive testing. Participants will complete an assessment at enrollment and once per year for the following 5 years. In addition to memory assessments at baseline and year 4, participants will have a brain MRI, OGTT A reliable study partner will need to attend the visits or be available via telephone to complete study interviews.
- Alzheimer's disease: This group will include 150 volunteers with mild stage Alzheimer's disease dementia. Participants will complete an assessment at enrollment and once per year for the following 5 years. In addition to memory assessments at baseline and year 4, participants will have a brain MRI, OGTT A reliable study partner will need to attend visits to complete study interviews.

SUMMARY:
Efforts to find treatments for AD have yielded only modest benefits, likely because longstanding AD pathological processes induce irreversible neurological compromise. These processes begin years before the onset of clinical symptoms. This possibility has been incorporated into a model describing stages of AD development, articulated by the NIA/Alzheimer's Association preclinical workgroup of which the Co-Director of the Kulynych Alzheimer's Research Center, Dr. Suzanne Craft, was a member. According to this model, the best hope for countermanding the effects of AD lies in intervening at the earliest possible point in the pathological cascade. There are several important ongoing efforts in adults with preclinical AD that directly target amyloid aggregation. Although this strategy addresses an important aspect of the AD pathological cascade, we believe that addressing metabolic dysfunction affecting glucose and insulin regulation offers a complementary approach, in that it may reduce amyloid burden and toxicity, while also directly enhancing synaptic health, brain metabolism, tau regulation and neurovascular function.

The purpose of the ADCC is to identify and characterize early risk factors that predict cognitive decline and dementia in asymptomatic adults and adults with early signs of cognitive impairment. The data obtained from this study, collected at enrollment and follow-up will allow us to examine disease trajectory in individuals with and without prediabetes and other measures of glucoregulatory dysfunction in this process. The enrollees, who will be well-characterized with regard to cognitive and metabolic status through ADCC assessments, will provide an important resource for other local (institution) and national investigations. Data collected from participants enrolled in the ADCC will be stored indefinitely for future investigations.

DETAILED DESCRIPTION:
The data and specimen repository of the ADCC study will provide a unified mechanism for cataloging and storing data that can be efficiently shared across studies. This repository will also allow for important collaborations with other Alzheimer's Disease Centers across the US that are performing similar investigations of adults at increased risk of dementia. Data sharing across multiple institutions and investigators will be critical to optimize speed of acquisition and standardization of outcomes that may ultimately lead to the development of innovative tools for early detection and new treatment strategies. The repository will include cognitive data, human specimen samples (blood, cerebrospinal fluid), medical and family history information, and neuroimaging data. Data collected from participants enrolled in the ADCC will be stored indefinitely for future investigations.

Participants will include adults at least 55 years old, with or without a cognitive deficit, who meet criteria for inclusion into one of the groups described below. Males and females will be equal to distribution in the Triad area population. Additional recruitment efforts targeting underserved communities will be used to increase representation of these adults in the study cohort beyond what is typical in other local and national studies of AD.

Eligible participants will have the option to participate in the core ADCC study and also in a biomarker-intensive substudy that will collect additional measurements of brain function and chemical markers of AD pathology. While all participants enrolled in the core ADCC study will receive brain magnetic resonance imaging (MRI). Those enrolled in the substudy will complete a lumbar puncture (LP) to permit quantification of AD biomarkers in cerebrospinal fluid (CSF). Participants enrolled in the substudy will be referred to as the Biomarker-Intensive Group, or ADCC-BIG.

At study entry, participants will meet inclusion criteria for membership in one of the groups that differ according to cognitive status and metabolic health (described below). Once enrolled, a change in cognitive or metabolic status will not affect eligibility to receive follow-up assessments as part of this study, although frequency of assessment may change (i.e., enrollees who progress to late-stage AD or type 2 diabetes will not be dis-enrolled). Eligible participants who choose to also enroll in ADCC-BIG must agree to complete the LP. If participants have screened or participated in another Kulynych Center study within the last 3 months, some data may be reused to avoid redundant data collection and reduce participant burden. This data may include specimen samples such as blood or CSF, cognitive testing data and MRI imaging data.

ELIGIBILITY:
Inclusion Criteria:

Group 1: Cognitively Normal (CN)

1. No subjective complaints of cognitive impairment
2. No cognitive impairment evident on formal testing interpreted by expert adjudication committee (typically, performance not worse than 1 SD below demographically relevant norms)
3. Clinical Dementia Rating (CDR) = 0 or 0.5
4. Normal glycemic control as indicated by American Diabetes Association (ADA) guidelines for normal 2 hour glycemic response to a glucose tolerance test (< 140 mg/dL).
5. Reliable collateral or study partner available to attend Visit 1 at a minimum

Group 2: Mild Cognitive Impairment (MCI)

1. Objective evidence of memory and/or executive function deficits on neuropsychological testing (typically 1.5 SD below demographically relevant norms)
2. CDR = 0 or 0.5
3. Reliable collateral or study partner

Group 3: Alzheimer's Disease (AD)

1. Diagnosis of probable mild AD, diagnosed with NIA-AA criteria, or mixed AD and vascular pathology as long as there is not a large vessel territory stroke, adjudicated by expert consensus panel.
2. Mini-Mental Status Exam (MMSE) score ≥ 10; CDR = ≥0.5
3. Normal glycemic control or prediabetes
4. Reliable collateral or study partner available to attend all visits

Exclusion Criteria:

1. Clinically significant abnormal labs
2. Significant neurologic disease that might affect cognition, other than AD, such as stroke, Parkinson's disease, multiple sclerosis, or recent severe head injury with loss of consciousness for more than 30 minutes within the last year, or with permanent neurologic sequelae
3. Clinically significant medical illness or organ failure as determined by study clinicians, including severe, uncontrolled cardiovascular disease, oxygen-treated chronic obstructive pulmonary disease, severe liver disease, Stage 4 chronic kidney disease or impending dialysis, active cancer, or other life-limiting condition with life expectancy less than 3 years
4. Current substance abuse or heavy alcohol consumption defined as >14 alcoholic drinks per week; or history of alcoholism or substance abuse within previous 10 years
5. Current poorly controlled depression or other psychiatric illness as determined by clinical judgement of study clinicians or neuropsychologists
6. Current use of anti-psychotic, benzodiazepines (PRN use <3 times per week is acceptable), anti-coagulants (for participants who will receive a lumbar puncture), strongly anticholinergic or sedative medications
7. Use of anticonvulsant for seizure disorder. (Use of anticonvulsant to treat other illnesses will be reviewed by the study MD and eligibility will be determined on a case by case basis.)
8. Current use of insulin
9. Brain MRI contraindications; including use of pacemakers, aneurysm clips, artificial heart valves, ear implants or metal/foreign objects in the eyes will be excluded from MRI
10. For participants completing any brain imaging protocol, inability to lie on the scanner bed for 40 minutes, or claustrophobia
11. For ADCC-BIG, significant obesity or a lower back condition that is likely to impede successful collection of CSF, as determined by study physician judgment
12. Other significant medical conditions at the investigators' discretion

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults, 55 years old and older, who have normal memory, mild memory impairment or AD. All subjects will be in reasonably good health with no significant medical illness that may contribute to memory decline other than MCI or probable AD.
Sampling Method: Probability Sample
Enrollment: 850 (Estimated)
Dates: Start 2014-01 (Actual); Primary Completion 2030-01 (Estimated); Study Completion 2031-01 (Estimated)

PRIMARY OUTCOMES:
Change in performance on cognitive measures. | 5 years
  Cognitive measure such as memory, verbal fluency and executive function will be assessed annually, either by phone or in person depending on group.

SECONDARY OUTCOMES:
Change in biomarker levels in cerebrospinal fluid (CSF). | 5 years
  Biomarkers associated with Alzheimer's will be measured in participants who agree to participate in the Biomarker-Intensive Group.
Change in brain volumes on magnetic resonance imaging (MRI). | 5 years
  MRI measures of brain volumes by region of interest, such as hippocampus, will be assessed during the baseline visit and again 3 years later (approximately week 156).

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Williamson, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Health, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
The ADCC is an observational study that will collect and store data at study entry and longitudinally for use in future studies. As part of the ADCC, the investigator will ask permission to store biological samples (blood, cerebrospinal fluid), as well as cognitive and medical data (neuroimaging, cognitive status, metabolic function markers, and family history information) indefinitely for future analyses. The Wake ADCC is part of a National collection of ADCCs funded by the NIA and as such, all centers contribute data to a central repository (National Alzheimer's Coordinating Center (NACC) at University of Washington). Participants will consent to have their de-identified data sent to the NACC.